CLINICAL TRIAL: NCT00842920
Title: Randomized Controlled Trial of Simvastatin in Amnestic MCI Patients
Brief Title: Trial of Simvastatin in Amnestic Mild Cognitive Impairment (MCI) Patients
Acronym: SIMaMCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Isabella Heuser, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT 2008-002226-11; BMBF grant, 01KG0822
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment
Keywords: amnestic MCI
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo or 20 mg Simvastatin (stratified by prior use of statins)
  Interventions: Drug: Placebo
- Simvastatin 60 mg (Experimental): Simvastatin 60 mg once daily
  Interventions: Drug: Simvastatin 60 mg
- Simvastatin 20 mg (Experimental): Simvastatin 20 mg once daily
  Interventions: Drug: Simvastatin 20 mg

INTERVENTIONS:
Drug: Simvastatin 60 mg — 60 mg once daily
  Arms: Simvastatin 60 mg
Drug: Placebo — one tablet once daily
  Arms: Placebo
Drug: Simvastatin 20 mg — 20 mg once daily
  Arms: Simvastatin 20 mg

SUMMARY:
Probands with MCI are at high risk to develop Alzheimer´s dementia (AD). Simvastatin may lower the production of Amyloid, a hallmark of AD in the brain. The primary hypothesis of the study is that 60 mg Simvastatin significantly reduces the Clinical Dementia Rating -Sum of boxes (CDR-SOB) in individuals with MCI as compared to MCI receiving placebo or 20 mg Simvastatin

DETAILED DESCRIPTION:
This is a national multicenter, double-blind, randomized placebo-controlled trial allowing for a minimum follow-up time of 24 months in conversion-free patients. Randomization will be stratified by prior use of statins.

The two strata are:

1. "no-statins": patients without treatment with a statins and no indication for treatment (according to the guidelines of the German Society of Cardiology for the primary prevention of cardiovascular disease); patients will be randomly assigned to one of 2 treatment (1) Simvastatin (60 mg) one tablet/day (2) Placebo one tablet/day.
2. "low-statins": patients treated with low doses of Statins; patients will be randomly assigned to one of 2 treatment (1) Simvastatin (60 mg) one tablet/day (2) 20 mg Simvastatin one tablet/day.

ELIGIBILITY:
Inclusion Criteria:

1. Self and informant report of gradually increasing memory impairment for at least six months.
2. Objective memory impairment
3. Intact basic activities of daily living
4. Preserved general cognitive function, not demented
5. Absence of a detectable cause of memory disorder
6. Age 55 to 90.
7. Females without childbearing potential
8. A total cholesterol ≥90 mg/dl
9. LDL-cholesterol ≥ 160 mg/dl and ≤ 3 risk factors or ≥ 190 mg/dl and ≤ 2 risk factors including age
10. Informed consent (according german medicinal products act, AMG §40 (1) 3b)
11. No participation in other clinical trials 2 months before and after participation in this study
12. Probands should only recruited for the clinical trial, when they are able to perform the informed consent; due to worsening of "memory function" in the course of the clinical trial, probands should not longer participate the clinical trial, when they is evidence, that participants were not longer able to give full informed consent.

Exclusion Criteria:

1. Hypersensitivity against Simvastatin, active liver disease or lasting increase of serum transaminases for unclear reason
2. Unstable medical, neurological or psychiatric disease
3. Lack of a spouse or a close relative
4. Use of a registered anti-dementia drug or a nootropic
5. Chronic use of anti-inflammatory drugs
6. History of stroke or myocardial infarction
7. LDL-cholesterol 130-160 mg/dl and > 3 risk factors or 160-190 mg/dl and > 2 risk factors including age.
8. LDL-cholesterol >190 mg/dl
9. Comedication with Diltiazem, Verapamil, Amiodarone, Itraconazole, Ketoconazole, Erythromycin, Clarithromycin, Telithromycin, Ciclosporin, Gemfibrozil, Nefazodone, HIV-protease inhibitors, Benzodiazepines, Tricyclic antipsychotics or other anticholinergic drugs
10. Comedication of other statins in high doses; low doses equivalent to 20 mg Simvastatin are allowed if taken for max. 2 years before randomization

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2008-12 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in CDR-SOB at 24 months of treatment | 24 month
  Clinical dementia rating - sum of boxes

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) score | 24 month
Change in Free and Cued Selective Reminding Test (FCSRT) score | 24 month
Length of conversion-free interval, starting at the time of randomization, with conversion being defined as an increase of the CDR score beyond 0.5 | 24 months

OTHER OUTCOMES:
Change in CDR-SOB at Long-Term Follow-Up | 2-11 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Heuser, MD, PhD, Principal Investigator — Charité-CBF; Lutz Frölich, MD, Principal Investigator — CIMH Mannheim
Locations (13):
- Germany (13):
  - Department of Psychiatry and Psychotherapy, Charité-CBF, Berlin
  - Department of Psychiatry and Psychotherapy, University Bonn, Bonn
  - Department of Psychiatry and Psychotherapy, University Erlangen, Erlangen
  - Department of Psychiatry and Psychotherapy, Johann Wolfgang Goethe-University, Frankfurt am Main
  - Center for Geriatrics and Gerontology, University Freiburg, Freiburg im Breisgau
  - Department of Psychiatry and Psychotherapy, Medical University Goettingen, Göttingen
  - Department for Psychiatry, Psychotherapy and Psychosomatic; Martin-Luther-University Halle-Wittenberg, Halle
  - Department of Psychiatry, University Hospital Heidelberg, Heidelberg
  - Department of Gerontopsychiatry, Central Institut of Mental Health, University Heidelberg, Mannheim
  - Department of Psychiatry and Psychotherapy, LMU I, Munich
  - Institute for Stroke and Dementia Research, LMU, Munich
  - Department of Psychiatry and Psychotherapy, University Rostock, Rostock
  - Neurologische Universitätsklinik Ulm, Ulm